CLINICAL TRIAL: NCT05364593
Title: Evaluating Point-of-care Ultrasound to Improve Tuberculosis Diagnosis in Children
Brief Title: Evaluation of Point-of-care Ultrasound in Children From 6 Months to 15 Years With Presumptive Tuberculosis
Status: Completed | Type: Observational
Sponsor: Medecins Sans Frontieres, Spain (Other)
Responsible Party: Principal Investigator, Laura Moreto, Principal Investigator, Medecins Sans Frontieres, Spain
Other Study IDs: MSF18116
Record Dates: First submitted 2022-04-26; First posted 2022-05-06 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Point of care ultrasound; FASH
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diagnosis of tuberculosis (TB) in children is particularly challenging in low and middle-income countries (LMIC), and a high number of children remain undiagnosed and untreated. A delay in diagnosis can lead to an increase in preventable morbidity and mortality. Point-of-care ultrasound (POCUS) is a bedside, non-invasive, inexpensive imaging tool, and TB-focused POCUS has been used and validated for adults with HIV. This study aims to describe the TB-focused POCUS findings for children with presumptive TB aged between 6 months and 15 years old, and to stratify the results per HIV, nutritional status and age. This is a Médecins Sans Frontières (MSF) multicentric study which takes place in Guinea Bissau and South Sudan.

DETAILED DESCRIPTION:
This study has as main objective to describe the findings obtained by POCUS methodology for pulmonary and extra-pulmonary tuberculosis in children per TB category. As secondary objectives: 1)To establish the sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of POCUS positive (any of 8 pre-established sonographic signs) as a composite against a composite reference of the final diagnosis (confirmed TB, unconfirmed TB or unlikely TB). 2)To describe the sonographic signs according to HIV status (positive, negative) and to nutritional status (SAM or not SAM). 3)To determine the proportion of children with improvement / resolution of sonographic signs and the proportion without improvement of sonographic signs at 2 months of follow-up in children with and without TB. 4)To describe operational aspects of POCUS: compliance with POCUS examination; quality of POCUS; duration of POCUS; mean time to definitive diagnostic in POCUS positive results compared to POCUS negative results; proportion of children who started TB treatment on basis of POCUS positive results.

This is a multicentric study in 2 different sites: Malakal (South Sudan) and Bissau (Guinea Bissau). The methodology for the evaluation of POCUS for the diagnosis of TB in children will be longitudinal case series with diagnostic test evaluation.

Study participants: The research population are children with presumptive TB in Malakal (town and POC hospitals) or in Bissau (Simão Mendes National Hospital).

Case with diagnosis of tuberculosis:

* Confirmed TB: patients with Xpert MTB/RIF positive (or TB culture positive when available) in a respiratory sample (pulmonary TB) or in other sample, such as CSF, lymph node or other tissue/liquid (extra pulmonary TB); TB LAM positive in HIV-infected patients.
* Unconfirmed TB: no microbiological confirmation but clinical diagnosis of TB and started on anti TB treatment (as established in Appendix 4).
* Unlikely TB: good response to other treatments (antibiotic, nutritional support, etc.) and no suggestive symptoms after 1 week of admission.

Identification of participants:

Eligible children will be identified upon admission to paediatric ward, ITFC, PICU/NICU (only in Bissau) or as suggestive cases in OPD. The identification of suspected TB cases will be mainly based on clinical criteria. A diagnostic algorithm (Appendix 4) will be applied to all suspected cases. The populations of interest for this study are hospitalized children, severely malnourished (SAM) and HIV positive or exposed children.

All TB cases (confirmed or unconfirmed) will be enrolled in TB care in MSF program (Malakal) or MoH program (Bissau). MSF will ensure that all patients to be started on adequate weight-based dose fix combinations and followed up during the length of treatment. All children diagnosed of DRTB will be initiated on DRTB treatment regimen according to national recommendation.

All patients included in the study (including those with unlikely TB) will provide telephone number (if available) and address. Whenever possible and if accepted by parent or guardian, a community health worker (CHW) will accompany the patient home after discharge. This CHW will be responsible for tracing the patients not attending the follow-up appointment. The CHWs are part of the Health Promotion / Community Engagement team and routinely involved in tracing of defaulters, including HIV/TB patients.

Safety Considerations : There are safety considerations related to infection control of TB, even if children are only considered contagious after they acquire the capacity of expectorating (> 8 years old). For older children, isolation procedures for coughing patients, as well as protection measures for medical staff, need to be implemented. Lab staff needs to wear respirator and gloves when manipulating samples for Xpert MTB/RIF. Safety procedures related to Xpert MTB/RIF need to be in place.

Diagnostic procedures are routinely done in all children with suspected TB (on not specifically for the study). Gastric lavage and naso-pharyngeal aspirate can be uncomfortable. For gastric lavage, there's a small risk of spasms of vocal cords, tube entering in the airway instead of the oesophagus, minor bleeding or aspiration pneumonia. Regarding naso-pharyngeal aspirate, the actual risks for participants are still smaller; it can cause nausea or local annoyance. Lymph node puncture is a routine procedure as well and is only performed in palpable lymph nodes (≥ 2 cm). The risks are small and can comprise blood vessel punction or accidental exposure to blood for the staff. All three are common procedures which will only be performed by trained staff. Any possible complication will be treated by MSF. No specific additional safety considerations related to POCUS.

Data Management and Analysis: The number of children tested by the program for suspected tuberculosis, the number of eligible children and the number of cases included in the study during the recruitment period will be noted. The number of parent or guardian of eligible children who refuse their participation will also be registered. Demographic, clinical and diagnostic characteristics at baseline and during patient follow-up under the program will also be recorded.

Data will be collected in the files by the study team members. Data will be coded and entered into a RedCap database and analysed with SPSS software. Continuous variables (e.g. age, distance) will be summarized using mean and standard deviation or median and interquartile range as appropriate and may also be expressed as ordinal categories with frequencies; frequencies will be reported with corresponding 95% confidence intervals. The main outcome of interest for POCUS study is to describe the findings obtained by POCUS methodology for pulmonary and extra pulmonary tuberculosis in children.

Bivariate analysis is planned for TB (confirmed and unconfirmed) vs unlikely TB, HIV positive vs. HIV negative, and for SAM vs. not SAM. Children with HIV and SAM will be considered as a confounder. Comparisons of these categorical variables across groups will use Chi-squared or Fisher's exact test. All estimates will be presented with respective 95% confidence intervals. Cohen's kappa coefficient will be used to determine the inter reader agreement of TB-focused POCUS positive, negative and per sign between the operator and second reader, and third reader in case of disagreement.

The number of children screened for suspected tuberculosis, the number of eligible children and the number of cases included in the study during the recruitment period will be noted. The number of parents or guardians of eligible children who refuse their participation will also be registered. Demographic, clinical and diagnostic characteristics at baseline and during patient follow-up under the program will also be recorded. Data analysis of the study will be conducted by the Epidemiologist/Statistician involved in the study, in collaboration with the PI.

Ethical Considerations:

The study will be conducted in accordance with the Declaration of Helsinki on Ethical Principles of Medical Research on Human Subjects, and in accordance with the rules of the National Ethics Committee of South Sudan and Guinea Bissau. The protocol will be submitted for approval to the National Committee for Ethics of South Sudan and Guinea Bissau, and the MSF Ethics Committee.

Informed consent: Participation in the study is on a voluntary basis and requires prior informed consent. Trained staff will provide eligible parents or guardians with detailed information on the study's objectives and procedures, as well as a clear explanation of the risks and benefits of participation. A written information sheet will be given to the parents or guardians, in English or in local language (appendix 1). The study staff will assist the parents or guardians on all the points indicated in the form and answer all the questions. If the parent or guardian is not able to read the information sheet, staff should read it aloud.

All children will be briefed on the study and the information will be adjusted to the age range and an assent process will take place for children older than 10 years old, but following national legislature, the consent must be signed by an adult. All questions will be answered by medical staff responsible for the study.

Parents or guardians agreeing to have their child participating in the study will need to sign an informed consent, which will also be signed by the study staff. For illiterate parents or guardians, a witness who can read and write, designated by the parent or guardian himself and who will not be a staff member of the study, will be present throughout the information process and will co-sign the form to confirm that the parents or guardians has understood and willingly accepts participation in the study.

The process of informed consent will be done in an area of the clinic that offers enough privacy to make a voluntary decision without constraint. Parents or guardians will be explicitly informed that they have the right to refuse participation or withdraw from the study at any time during the research. Copies of both forms (ie. the study information sheet and informed consent, in English or in the local language) will be given to the parents or guardians.

Confidentiality: All information collected during the study will be recorded and identified by a specifically assigned number for the study and the number assigned routinely for the program. Patient or parents or guardians names will not be recorded in the study form or electronic databases. Access to the study information (in paper or electronic format) is restricted to authorized staff.

Home visits are part of the regular work of CHWs, who have specifically been trained for this task. To guarantee confidentiality, they are not informed about the reason of the visit and just deliver a request to attend the clinic as soon as possible. This information has been shared with the local authorities and is routinely explained to all patients prior to asking for consent for home visits.

Informed consent forms will be kept in a secure and confidential place in a locked cabinet by the study coordinator throughout the study. The consent forms will be archived for a minimum of 5 years after the end of the research, in a secure and locked archive by the investigator at MSF OCBA, in Barcelona. After this period, all documents will be destroyed. If the Ministry of Health requests to archive copies of the informed consents, they will be given at the end of the research study.

ELIGIBILITY:
Inclusion Criteria:

* Any child from 6 months of life to 15 years old
* Presumptive TB according to diagnostic criteria
* Informed consent provided by legal responsible or companion

Exclusion Criteria:

* Patients who have received TB treatment for > 1 day in the last 3 months
* Informed consent not provided by legal responsible or companion

Ages: 6 Months to 15 Years | Sex: All
Age Groups: Child
Study Population: The study population are children with presumptive TB in Malakal (South Sudan) and at Simão Mendes National Hospital in Bissau (Guinea-Bissau).
Sampling Method: Non-Probability Sample
Enrollment: 576 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
To describe the sonographic findings obtained by TB-focused POCUS methodology | At baseline
  To describe the sonographic findings obtained by TB-focused POCUS methodology for pulmonary and extra-pulmonary tuberculosis in children per TB category

SECONDARY OUTCOMES:
To establish the sensitivity, specificity, positive predictive value and negative predictive value of POCUS positive as a composite against a composite reference of the final diagnosis | At baseline
  To establish the sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of POCUS positive (any of 8 pre-established sonographic signs) as a composite against a composite reference of the final diagnosis (confirmed TB, unconfirmed TB or unlikely TB)
To describe the sonographic signs according to HIV status (positive, negative) | At baseline
  To describe the sonographic signs according to HIV status (positive, negative)
To describe the sonographic signs according to nutritional status (severe acute malnutrition (SAM) or not SAM) | At baseline
  To describe the sonographic signs according to nutritional status (SAM or not SAM)
To determine the proportion of children with improvement / resolution of sonographic signs and the proportion without improvement of sonographic signs at 2 months of follow-up in children with and without TB | At 2 months
  To determine the proportion of children with improvement / resolution of sonographic signs and the proportion without improvement of sonographic signs at 2 months of follow-up in children with and without TB
To describe operational aspects of POCUS: compliance | At baseline
  To describe operational aspects of POCUS: compliance with POCUS examination
To describe operational aspects of POCUS: duration of POCUS | At baseline
  To describe operational aspects of POCUS: duration in minutes of POCUS procedure
To describe operational aspects of POCUS: mean time to diagnosis | At baseline
  To describe operational aspects of POCUS: mean time to definitive diagnostic in POCUS positive results compared to POCUS negative results

CONTACTS AND LOCATIONS:
Overall Officials: Laura Moretó, MD, MIH, Principal Investigator — MSF OCBA; Sabine Belard, MD, PhD, Principal Investigator — University Hospital Tuebingen
Locations (2):
- Simao Mendes Hospital, Bissau, Guinea-Bissau
- Malakal hospital, Malakal, Upper Nile, South Sudan

IPD SHARING:
Plan to Share IPD: Undecided
We have not yet decided to make the IPD available for other researchers.

REFERENCES:
- [Background] Mwangwa F, Chamie G, Kwarisiima D, Ayieko J, Owaraganise A, Ruel TD, Plenty A, Tram KH, Clark TD, Cohen CR, Bukusi EA, Petersen M, Kamya MR, Charlebois ED, Havlir DV, Marquez C. Gaps in the Child Tuberculosis Care Cascade in 32 Rural Communities in Uganda and Kenya. J Clin Tuberc Other Mycobact Dis. 2017 Dec;9:24-29. doi: 10.1016/j.jctube.2017.10.003. PMID 29291251
- [Background] Chisti MJ, Ahmed T, Pietroni MA, Faruque AS, Ashraf H, Bardhan PK, Hossain I, Das SK, Salam MA. Pulmonary tuberculosis in severely-malnourished or HIV-infected children with pneumonia: a review. J Health Popul Nutr. 2013 Sep;31(3):308-13. doi: 10.3329/jhpn.v31i3.16516. PMID 24288943
- [Background] Jaganath D, Mupere E. Childhood tuberculosis and malnutrition. J Infect Dis. 2012 Dec 15;206(12):1809-15. doi: 10.1093/infdis/jis608. Epub 2012 Oct 2. PMID 23033147
- [Background] Graham SM, Ahmed T, Amanullah F, Browning R, Cardenas V, Casenghi M, Cuevas LE, Gale M, Gie RP, Grzemska M, Handelsman E, Hatherill M, Hesseling AC, Jean-Philippe P, Kampmann B, Kabra SK, Lienhardt C, Lighter-Fisher J, Madhi S, Makhene M, Marais BJ, McNeeley DF, Menzies H, Mitchell C, Modi S, Mofenson L, Musoke P, Nachman S, Powell C, Rigaud M, Rouzier V, Starke JR, Swaminathan S, Wingfield C. Evaluation of tuberculosis diagnostics in children: 1. Proposed clinical case definitions for classification of intrathoracic tuberculosis disease. Consensus from an expert panel. J Infect Dis. 2012 May 15;205 Suppl 2(Suppl 2):S199-208. doi: 10.1093/infdis/jis008. Epub 2012 Mar 22. PMID 22448023
- [Background] Belard S, Tamarozzi F, Bustinduy AL, Wallrauch C, Grobusch MP, Kuhn W, Brunetti E, Joekes E, Heller T. Point-of-Care Ultrasound Assessment of Tropical Infectious Diseases--A Review of Applications and Perspectives. Am J Trop Med Hyg. 2016 Jan;94(1):8-21. doi: 10.4269/ajtmh.15-0421. Epub 2015 Sep 28. PMID 26416111
- [Background] Bobbio F, Di Gennaro F, Marotta C, Kok J, Akec G, Norbis L, Monno L, Saracino A, Mazzucco W, Lunardi M. Focused ultrasound to diagnose HIV-associated tuberculosis (FASH) in the extremely resource-limited setting of South Sudan: a cross-sectional study. BMJ Open. 2019 Apr 2;9(4):e027179. doi: 10.1136/bmjopen-2018-027179. PMID 30944140
- [Background] Heller T, Wallrauch C, Goblirsch S, Brunetti E. Focused assessment with sonography for HIV-associated tuberculosis (FASH): a short protocol and a pictorial review. Crit Ultrasound J. 2012 Nov 21;4(1):21. doi: 10.1186/2036-7902-4-21. PMID 23171481
- [Background] Heller T, Goblirsch S, Bahlas S, Ahmed M, Giordani MT, Wallrauch C, Brunetti E. Diagnostic value of FASH ultrasound and chest X-ray in HIV-co-infected patients with abdominal tuberculosis. Int J Tuberc Lung Dis. 2013 Mar;17(3):342-4. doi: 10.5588/ijtld.12.0679. Epub 2013 Jan 14. PMID 23321507
- [Background] Weber SF, Saravu K, Heller T, Kadavigere R, Vishwanath S, Gehring S, Belard S, And Pocus Eti Study Group. Point-of-Care Ultrasound for Extrapulmonary Tuberculosis in India: A Prospective Cohort Study in HIV-Positive and HIV-Negative Presumptive Tuberculosis Patients. Am J Trop Med Hyg. 2018 Jan;98(1):266-273. doi: 10.4269/ajtmh.17-0486. PMID 29141727
- [Background] Heller T, Mtemang'ombe EA, Huson MA, Heuvelings CC, Belard S, Janssen S, Phiri S, Grobusch MP. Ultrasound for patients in a high HIV/tuberculosis prevalence setting: a needs assessment and review of focused applications for Sub-Saharan Africa. Int J Infect Dis. 2017 Mar;56:229-236. doi: 10.1016/j.ijid.2016.11.001. Epub 2016 Nov 9. PMID 27836795
- [Background] Griesel R, Cohen K, Mendelson M, Maartens G. Abdominal Ultrasound for the Diagnosis of Tuberculosis Among Human Immunodeficiency Virus-Positive Inpatients With World Health Organization Danger Signs. Open Forum Infect Dis. 2019 Apr 7;6(4):ofz094. doi: 10.1093/ofid/ofz094. eCollection 2019 Apr. PMID 31011588
- [Background] Kahn D, Pool KL, Phiri L, Chibwana F, Schwab K, Longwe L, Banda BA, Gama K, Chimombo M, Chipungu C, Grotts J, Schooley A, Hoffman RM. Diagnostic Utility and Impact on Clinical Decision Making of Focused Assessment With Sonography for HIV-Associated Tuberculosis in Malawi: A Prospective Cohort Study. Glob Health Sci Pract. 2020 Mar 31;8(1):28-37. doi: 10.9745/GHSP-D-19-00251. Print 2020 Mar 30. PMID 32041772
- [Background] Heuvelings CC, Belard S, Andronikou S, Jamieson-Luff N, Grobusch MP, Zar HJ. Chest ultrasound findings in children with suspected pulmonary tuberculosis. Pediatr Pulmonol. 2019 Apr;54(4):463-470. doi: 10.1002/ppul.24230. Epub 2019 Jan 11. PMID 30632712
- [Background] Belard S, Heller T, Orie V, Heuvelings CC, Bateman L, Workman L, Grobusch MP, Zar HJ. Sonographic Findings of Abdominal Tuberculosis in Children With Pulmonary Tuberculosis. Pediatr Infect Dis J. 2017 Dec;36(12):1224-1226. doi: 10.1097/INF.0000000000001590. PMID 28333710
- [Background] Belard S, Heller T, Grobusch MP, Zar HJ. Point-of-care ultrasound: a simple protocol to improve diagnosis of childhood tuberculosis. Pediatr Radiol. 2014 Jun;44(6):679-80. doi: 10.1007/s00247-014-2971-7. Epub 2014 May 23. No abstract available. PMID 24854937
- [Background] Belard S, Heuvelings CC, Banderker E, Bateman L, Heller T, Andronikou S, Workman L, Grobusch MP, Zar HJ. Utility of Point-of-care Ultrasound in Children With Pulmonary Tuberculosis. Pediatr Infect Dis J. 2018 Jul;37(7):637-642. doi: 10.1097/INF.0000000000001872. PMID 29278611
- [Background] Abrokwa SK, Ruby LC, Heuvelings CC, Belard S. Task shifting for point of care ultrasound in primary healthcare in low- and middle-income countries-a systematic review. EClinicalMedicine. 2022 Mar 6;45:101333. doi: 10.1016/j.eclinm.2022.101333. eCollection 2022 Mar. PMID 35284806
- [Derived] Moreto-Planas L, Sagrado MJ, Mahajan R, Gallo J, Biague E, Goncalves R, Nuozzi P, Rocaspana M, Fonseca JV, Medina C, Camara M, Nadimpalli A, Alonso B, Llosa AE, Heuvelings L, Burza S, Molina I, Ruby LC, Stratta E, Belard S. Point-of-care ultrasound for tuberculosis diagnosis in children: a Medecins Sans Frontieres cross-sectional study in Guinea-Bissau. BMJ Open. 2023 May 19;13(5):e066937. doi: 10.1136/bmjopen-2022-066937. PMID 37208138

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT05364593/Prot_ICF_000.pdf